CLINICAL TRIAL: NCT02326194
Title: A Phase 1 Double-blind, Dose-escalation, Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of the Ebola Adenovirus Vector Vaccine (Ad5-EBOV) in Healthy Adults in China
Brief Title: A Phase I Clinical Trial to Evaluate the Ebola Adenovirus Vector Vaccine (Ad5-EBOV) in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Beijing Institute of Biotechnology (Other); Tianjin Cansino Biotechnology Inc (Industry)
Responsible Party: Principal Investigator, Fengcai Zhu, Jiangsu Province Centers for Disease Control and Prevention, Jiangsu Province Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT020
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Ebola Virus Disease
Keywords: Safety,immunogenicity,Ebola
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo group (one shot) (Placebo Comparator): one dose
  Interventions: Biological: placebo (one dose)
- Placebo group (two shots) (Placebo Comparator): two doses, with one dose to each arm at a same time.
  Interventions: Biological: placebo (two doses)
- Low dose vaccine group (Experimental): one dose, low dose Ebola Zaire vaccine (Ad5-EBOV)
  Interventions: Biological: Low dose Ebola Zaire vaccine (Ad5-EBOV)
- High dose vaccine group (Experimental): two doses, high dose, with one dose to each arm at a same time
  Interventions: Biological: High dose Ebola Zaire vaccine (Ad5-EBOV)

INTERVENTIONS:
Biological: Low dose Ebola Zaire vaccine (Ad5-EBOV) — one dose, Low dose Ebola Zaire vaccine (Ad5-EBOV)
  Arms: Low dose vaccine group
Biological: High dose Ebola Zaire vaccine (Ad5-EBOV) — two doses, High dose Ebola Zaire vaccine (Ad5-EBOV), with one dose to each arm at a same time.
  Arms: High dose vaccine group
Biological: placebo (one dose) — placebo, one doses
  Arms: Placebo group (one shot)
Biological: placebo (two doses) — placebo, two doses, with one dose to each arm at a same time.
  Arms: Placebo group (two shots)

SUMMARY:
Since its first outbreak occurred in 1976, Zaire Ebola virus have been associated with 14 outbreaks reported up to 2014. The Zaire Ebola virus in 2014 causing the most serious outbreak was considered to be a new epidemic strain, with GP homology of the gene was only 97.6%, compared to the GP gene of the strain in 1976. This investigational Ad5-EBOV vaccine was developed according to the 2014 epidemic Zaire strain and formulated as freeze-dry products which could be stored at 4℃.

This is a single center, double-blind, placebo control, dose-escalation phase 1 clinical trial. This study will determine the safety and side-effect profile, and immunogenicity of an investigational Ad5-EBOV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years.
* Able to understand the content of informed consent and willing to sign the informed consent
* Able and willing to complete all the secluded study process during the whole study follow-up period (about 6 months).
* A body mass index (BMI) <35
* Hemoglobin 110-150g/L for female, and 120-160g/L for male.
* White blood cells (WBC) 4.0-10.0×109 cells/L
* Total lymphocyte Count 0.8-4.5×109 cells/L
* Platelets 100-300×109 cells/L
* Alanine aminotransferase (ALT) 0-40U/L
* Serum creatinine 44-106μmol/L
* Partial thromboplastin time (PTT) 20-40 seconds
* Prothrombin time (PT) 10-14 seconds
* Negative in HIV diagnostic blood test
* Axillary temperature ≤37.0°C on the day of enrollment
* General good health as established by medical history and physical examination.

Exclusion Criteria:

* Family history of seizure, epilepsy, brain or mental disease
* Subject that has a medical history of any of the following: allergic history of any vaccination or drugs, or allergic to any ingredient of the Ad5-EBOV vaccine, such as mannitol
* Woman who is pregnant, breast-feeding or positive in β-HCG (human chorionic gonadotropin) pregnancy test (urine) on day of enrollment, or become pregnant during the next 6 months
* Any acute fever disease or infections in last 7 days
* Major congenital defects or not well-controlled chronic illness, such as asthma, diabetes, or thyroid disease
* Hereditary angioneurotic edema or acquired angioneurotic edema
* Urticaria in last one year
* Asplenia or functional asplenia
* Platelet disorder or other bleeding disorder may cause injection contraindication
* Faint at the sight of blood or needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylaxis treatment, cytotoxic treatment in last 6 months
* Prior administration of blood products in last 4 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine in last 1 month
* Prior administration of inactivated vaccine in last 14 days
* Current anti-tuberculosis prophylaxis or therapy
* Any condition that in the opinion of the investigators may interfere with the evaluation of study objectives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse reactions after vaccination. | within 7 days after the vaccination
  Occurrence of adverse reactions within 7 days after vaccination with the Ebola Zaire vaccine (Ad5-EBOV).
Specific anti-EBOV antibody responses to the Ebola Zaire vaccine (Ad5-EBOV). | 28 days after the vaccination
  Specific anti-EBOV antibody responses to the Ebola Zaire vaccine (Ad5-EBOV) as measured by ELISA.
Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV). | 28 days after the vaccination
  Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV) as measured by intracellular cytokine staining assays (ICS)

SECONDARY OUTCOMES:
Occurrence of adverse events after the vaccination. | within 28 days after the vaccination
  Occurrence of adverse events within 28 days after vaccination with the Ebola Zaire vaccine (Ad5-EBOV).
Changes of the laboratory examinations after vaccination. | day 0-28 after the vaccination
  Changes of the laboratory examinations after vaccination with the Ebola Zaire vaccine (Ad5-EBOV) on day 3, 14 and 28.
Occurrence of serious adverse events after the vaccination. | within 6 months after the vaccination
  Occurrence of serious adverse events within 6 months after the vaccination with the Ebola Zaire vaccine (Ad5-EBOV).
Specific anti-EBOV antibody responses to the Ebola Zaire vaccine (Ad5-EBOV). | 168 days after the vaccination
  Specific anti-EBOV antibody responses to the Ebola Zaire vaccine (Ad5-EBOV) at day 168 as measured by ELISA.
Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV). | 168 days after the vaccination
  Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV) at day 168 as measured by intracellular cytokine staining assays (ICS).
Anti-adenovirus neutralizing antibody responses to the Ebola Zaire vaccine (Ad5-EBOV). | 168 days after the vaccination
  Anti-adenovirus neutralizing antibody responses to the Ebola Zaire vaccine (Ad5-EBOV) at day 168.

OTHER OUTCOMES:
Changes of the laboratory examinations after vaccination. | day 168 after the vaccination
  Changes of the laboratory examinations after vaccination with the Ebola Zaire vaccine (Ad5-EBOV) at day 168.
Specific anti-EBOV antibody responses to the Ebola Zaire vaccine (Ad5-EBOV). | 3-112 days after the vaccination
  Specific anti-EBOV antibody responses to the Ebola Zaire vaccine (Ad5-EBOV) at day 3, 7, 14, 56 and 112 as measured by ELISA.
Anti-adenovirus neutralizing antibody responses to the Ebola Zaire vaccine (Ad5-EBOV). | 3-56 days after the vaccination
  Anti-adenovirus neutralizing antibody responses to the Ebola Zaire vaccine (Ad5-EBOV) at day 3, 7, 14, 56 and 112.
Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV). | day 7-112 after the vaccination
  Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV) at day 7, 14, 56 and 112 as measured by intracellular cytokine staining assays (ICS).
Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV). | day 0-168 after the vaccination
  Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV) at day 0, 28 and 168 as measured by ELISpot.

CONTACTS AND LOCATIONS:
Locations (1):
- Phase 1 vaccine clinical trial center of Jiangsu Provincial Center for Disease Control and Prevention, Taizhou, Jiangsu, China

REFERENCES:
- [Derived] Li JX, Hou LH, Meng FY, Wu SP, Hu YM, Liang Q, Chu K, Zhang Z, Xu JJ, Tang R, Wang WJ, Liu P, Hu JL, Luo L, Jiang R, Zhu FC, Chen W. Immunity duration of a recombinant adenovirus type-5 vector-based Ebola vaccine and a homologous prime-boost immunisation in healthy adults in China: final report of a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Glob Health. 2017 Mar;5(3):e324-e334. doi: 10.1016/S2214-109X(16)30367-9. Epub 2016 Dec 23. PMID 28017642
- [Derived] Zhu FC, Hou LH, Li JX, Wu SP, Liu P, Zhang GR, Hu YM, Meng FY, Xu JJ, Tang R, Zhang JL, Wang WJ, Duan L, Chu K, Liang Q, Hu JL, Luo L, Zhu T, Wang JZ, Chen W. Safety and immunogenicity of a novel recombinant adenovirus type-5 vector-based Ebola vaccine in healthy adults in China: preliminary report of a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet. 2015 Jun 6;385(9984):2272-9. doi: 10.1016/S0140-6736(15)60553-0. Epub 2015 Mar 25. PMID 25817373